CLINICAL TRIAL: NCT04981756
Title: Primary Sclerosing Cholangitis in China: Epidemiology, Cascade and Treatment
Brief Title: PSC Clinical Epidemiology in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); Shanghai Suvalue Health Scientific Ltd. (Unknown); The First Hospital of Jilin University (Other); Beijing Ditan Hospital (Other); Tianjin Medical University General Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Hospital of Jilin University (Other); Hepatobiliary Disease Hospital of Jilin Province (Unknown); Lanzhou University Second Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Jidong Jia, Director of Liver Research Center, Beijing Friendship Hospital
Other Study IDs: IN-CN-428-5940
Record Dates: First submitted 2021-06-23; First posted 2021-07-29 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Epidemiology; Cascade; Treatment
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — This observational study does not have any intervention.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a rare disease but is increasingly reported in China (mainly in the Chinese language). However, most of the PSC literatures reported from China are case reports, small case series, and review articles. Up to now, there is no information on the epidemiology and disease burden of PSC in China. This study would use EMR/HIS and research databases to investigate the epidemiology, cascade, and treatment pattern of PSC in China.

DETAILED DESCRIPTION:
Identify the PSC cases diagnosed from the earliest date available to the present in the SuValue Research Database and the HIS/EMR from clinical sites through diagnostic ICD codes, laboratory, pathology, imaging, endoscopy, surgery, medication, hospitalization, and health outcomes.

Collect information on PSC cases' key demographic, the time of PSC diagnosis, hematological/biochemical variables (ALT, AST, ALP, GGT, ALP TBil, ALB), MRCP or ERCP or pathological report, IBD (UC or CD) symptoms, or colon, medication information, clinical outcomes (including cirrhosis, decompensated cirrhosis, death or liver transplantation) as well as current or past treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Retrospectively review PSC cases before April 1, 2002 will be identified by diagnostic codes from the International Classification of Diseases (ICD)-9, and for those after April 1, 2002, we used ICD-10.
2. We identified patients using an electronic search of SuValue Research Database and HIS of BFH-CMU and BYH-CMU using PSC related ICD codes (ICD-9: 576.1; ICD-10: K83.016/K83.016(China version)). To supplement the ICD search, an electronic keyword search for "primary sclerosing cholangitis" or "seclerosing cholangitis" was conducted on all radiology, endoscopy, pathology reports beginning on earliest date available in the database of SuValue Research Database and HIS of BFH-CMU and BYH-CMU. We reviewed the medical charts of identified patients and diagnostic criteria including cholestatic biochemistry (ALP, GGT elevations), and typical imaging (MRCP or ERCP) or pathological features, excluding other known etiology. For patients with multiple visits for PSC, we reviewed only the index visit. To ensure consistency, chart review was independently assessed by two hepatologists. Discrepancies in compliance were resolved by discussion between the two main reviewers. Any unresolved discrepancies were decided by a third expert hepatologist.

Exclusion Criteria:

1. The cases with secondary sclerosing cholangitis caused by cholelithiasis, IgG4 related disease, malignancy or other known etiologies.
2. The cases with missing key results on clinical, biochemical (ALP, GGT, bilirubin), radiological (MRCP or ERCP) or histological investigations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total number of subjects expected to be reviewed is 800. The subjects in this study will consist of two parts: identify PSC cases by retrospective review of an inter-regional database and retro-prospective review of EMR of two tertiary medical centers in Beijing.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of PSC | 7 years
  The crude prevalence of PSC patients
Crowd Distribution of PSC in China | 7 years
  Crowd distribution includes the age-specified/sex-specified distribution

SECONDARY OUTCOMES:
The positive rate of ANCA | 0 to 7 years
  The percentage of patients with anti-neutrophil cytoplasmic antibodies (ANCA) positive
Dynamic changes of aminotransferase | 0 to 7 years
  Dynamic changes of alanine aminotransferase (ALT) from year-0 to year-7
Dynamic changes of aspartate aminotransferase | 0 to 7 years
  Dynamic changes of aspartate aminotransferase (AST) from year-0 to year-7
Dynamic changes of alkaline phosphatase | 0 to 7 years
  Dynamic changes of alkaline phosphatase (ALP) from year-0 to year-7
Dynamic changes of gamma-glutamyl transpeptidase | 0 to 7 years
  Dynamic changes of gamma-glutamyl transpeptidase (GGT) from year-0 to year-7
Dynamic changes of serum total bilirubin | 0 to 7 years
  Dynamic changes of serum total bilirubin (TBIL) from year-0 to year-7
Dynamic changes of the radiological features measured by Magnetic Resonance Cholangiopancreatography (MRCP) or Encoscopic Retrograde Cholangio-Pancreatography (ERCP) | 0 to 7 years
  Dynamic changes of the radiological features at baseline and after 1, 3, 5, 7 years of treatment
Incidence of concomitant diseases | 0 to 7 years
  Concomitant diseases include IBD (UC or CD), AIH, PBC, cirrhosis, cholelithiasis or cholangiocarcinoma
Cumulative incidence of clinical outcomes | 0 to 7 years
  Cumulative incidence of liver decompensation (including ascites, hepatic encephalopathy, esophageal varices bleeding and Hepatocellular Carcinoma) , liver transplantation, cholangiocarcinoma and death
The medication information | 0 to 7 years
  Document medication information from year-0 to year-7

CONTACTS AND LOCATIONS:
Overall Officials: Jidong Jia, MD, PhD, Principal Investigator — Beijing Friendship Hospital, Capital Medical University, Beijing, China
Locations (3):
- China (3):
  - Beijing Friendship Hospital, Capital Medical Univeristy, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shanghai Suvalue Health Scientific Ltd., Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ponsioen CY, Lindor KD, Mehta R, Dimick-Santos L. Design and Endpoints for Clinical Trials in Primary Sclerosing Cholangitis. Hepatology. 2018 Sep;68(3):1174-1188. doi: 10.1002/hep.29882. Epub 2018 Aug 31. PMID 29574971
- [Background] Deneau M, Jensen MK, Holmen J, Williams MS, Book LS, Guthery SL. Primary sclerosing cholangitis, autoimmune hepatitis, and overlap in Utah children: epidemiology and natural history. Hepatology. 2013 Oct;58(4):1392-400. doi: 10.1002/hep.26454. Epub 2013 Aug 13. PMID 23686586
- [Background] Boonstra K, Weersma RK, van Erpecum KJ, Rauws EA, Spanier BW, Poen AC, van Nieuwkerk KM, Drenth JP, Witteman BJ, Tuynman HA, Naber AH, Kingma PJ, van Buuren HR, van Hoek B, Vleggaar FP, van Geloven N, Beuers U, Ponsioen CY; EpiPSCPBC Study Group. Population-based epidemiology, malignancy risk, and outcome of primary sclerosing cholangitis. Hepatology. 2013 Dec;58(6):2045-55. doi: 10.1002/hep.26565. Epub 2013 Oct 17. PMID 23775876
- [Background] Metcalf J, James O. The geoepidemiology of primary biliary cirrhosis. Semin Liver Dis. 1997 Feb;17(1):13-22. doi: 10.1055/s-2007-1007179. PMID 9089907
- [Background] Liu K, Wang R, Kariyawasam V, Wells M, Strasser SI, McCaughan G, Corte C, Leong RW. Epidemiology and outcomes of primary sclerosing cholangitis with and without inflammatory bowel disease in an Australian cohort. Liver Int. 2017 Mar;37(3):442-448. doi: 10.1111/liv.13328. Epub 2017 Jan 24. PMID 27891750
- [Background] Shen T, Liu Y, Shang J, Xie Q, Li J, Yan M, Xu J, Niu J, Liu J, Watkins PB, Aithal GP, Andrade RJ, Dou X, Yao L, Lv F, Wang Q, Li Y, Zhou X, Zhang Y, Zong P, Wan B, Zou Z, Yang D, Nie Y, Li D, Wang Y, Han X, Zhuang H, Mao Y, Chen C. Incidence and Etiology of Drug-Induced Liver Injury in Mainland China. Gastroenterology. 2019 Jun;156(8):2230-2241.e11. doi: 10.1053/j.gastro.2019.02.002. Epub 2019 Feb 8. PMID 30742832
- [Background] Colbaugh R, Glass K, Rudolf C, Tremblay Volv Global Lausanne Switzerland M. Learning to Identify Rare Disease Patients from Electronic Health Records. AMIA Annu Symp Proc. 2018 Dec 5;2018:340-347. eCollection 2018. PMID 30815073
- [Background] Sada Y, Hou J, Richardson P, El-Serag H, Davila J. Validation of Case Finding Algorithms for Hepatocellular Cancer From Administrative Data and Electronic Health Records Using Natural Language Processing. Med Care. 2016 Feb;54(2):e9-14. doi: 10.1097/MLR.0b013e3182a30373. PMID 23929403